CLINICAL TRIAL: NCT04723433
Title: Recovery of Ventilation After General Anesthesia for Robotic-assisted Laparoscopic Nephrectomy: The Effect of Conservative Versus Liberal Oxygen Supplementation - A Feasibility Study
Brief Title: Recovery of Ventilation After Anesthesia for Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, Professor, Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-59593
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Ventilatory Depression; Postoperative Respiratory Complication
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: In the post-anesthesia care unit (PACU), participants will be randomized to receive conservative (titrated to an SpO2 between 90 and 94%) versus liberal (titrated to SpO2 > 96%) oxygen supplementation, via a non-rebreather mask.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Conservative O2 Supplementation" (Experimental): Oxygen administration will titrated to a oxyhemoglobin saturation (SpO2) between 90 and 94%.
  Interventions: Other: Oxygen gas -Conservative
- "Liberal O2 Supplementation" (Active Comparator): Oxygen administration will titrated to an SpO2 > 96%.
  Interventions: Other: Oxygen gas -Liberal

INTERVENTIONS:
Other: Oxygen gas -Conservative — Oxygen administration will titrated to a oxyhemoglobin saturation (SpO2) between 90% and 94%.
  Arms: "Conservative O2 Supplementation"
Other: Oxygen gas -Liberal — Oxygen administration will titrated to a oxyhemoglobin saturation (SpO2) higher than 96%.
  Arms: "Liberal O2 Supplementation"

SUMMARY:
The purpose of this randomized, controlled feasibility investigation is to characterize pharmacologically induced ventilatory depression after anesthesia and examine how is affected by the amount of supplemental oxygen patients are receiving in the immediate postoperative period.

DETAILED DESCRIPTION:
The purpose of this study is characterize pharmacologically induced ventilatory depression after anesthesia and examine how is affected by the amount of supplemental oxygen patients are receiving in the immediate postoperative period, since hyperoxemia (ie., higher than necessary partial pressure of oxygen in the arterial blood) has been associated with ventilatory depression via suppression of the hypoxic ventilatory drive.

In this feasibility randomized controlled trial, the investigators plan to estimate and compare the cumulative segment of time during which the transcutaneous partial pressure of carbon dioxide will exceed an upper limit of 45 mmHg (i.e., TcPCO2 > 45 mmHg) for the 90-min-long post-anesthesia period, between the conventional (titrated to an oxygen saturation > 96%) and the conservative (titrated to O2 saturation 90 -94%) O2 supplementation interventions.

Hypothesis: Conservative use of O2 (titrated to an SpO2: 90 - 94%), will be associated with less hypoventilation (i.e., less time spent with an TcPCO2 > 45 mmHg) during recovery from general anesthesia, compared to liberal O2 supplementation (SpO2 > 96%).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Body mass index (BMI) less than 40 kg/m2
* Scheduled to undergo robotic-assisted radical laparoscopic nephrectomy.

Exclusion Criteria:

* Patients with a diagnosis of chronic obstructive pulmonary disorder (COPD), severe neurological, cardiopulmonary, psychiatric, or untreated thyroid disorder
* Chronic pain condition that is being treated with opioids
* Patients with a hematocrit lower than 30% at the end of surgery, or those with an excessive blood loss, requiring transfusion of blood products during their surgery, will be also excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Transcutaneous partial pressure of carbon dioxide (TcPCO2) | Ninety -minute period immediately post-anesthesia.
  The cumulative segment of time during which the transcutaneous partial pressure of carbon dioxide (TcPCO2: primary outcome) will exceed an upper limit of 45 mmHg (i.e., TcPCO2 > 45 mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doufas AG, Tian L, Kutscher S, Finnsson E, Agustsson JS, Chung BI, Panousis P. The effect of hyperoxia on ventilation during recovery from general anesthesia: A randomized pilot study for a parallel randomized controlled trial. J Clin Anesth. 2022 Dec;83:110982. doi: 10.1016/j.jclinane.2022.110982. Epub 2022 Oct 17. PMID 36265267